CLINICAL TRIAL: NCT05714657
Title: A Phase II Study of Shortened Course, Dose De-Intensified Adjuvant Radiotherapy Following Transoral Robotic Surgery (TORS) and Neck Dissection for HPV-Associated Oropharyngeal Squamous Cell Carcinoma
Brief Title: Shortened Course Adjuvant Radiotherapy Following TORS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 06322; 852738 (Other: University of Pennsylvania Institutional Review Board)
Record Dates: First submitted 2022-08-03; First posted 2023-02-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: HPV-Associated Oropharyngeal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Shortened Course Adjuvant Radiotherapy (Experimental): The volume treated to the regional lymphatics will be according to the characteristics of the primary site and involved lymph nodes. The dose of radiotherapy delivered will be 30 Gy, over the course of 10 treatments (5 daily treatments/week).
  Treatment of the primary tumor bed will be omitted in appropriate patients, as per the initial TORS de-intensification protocol. In patients requiring treatment of the primary site, reduced dose (30 Gy) will be delivered.
  Interventions: Radiation: Shortened Course Adjuvant Radiotherapy Following TORS

INTERVENTIONS:
Radiation: Shortened Course Adjuvant Radiotherapy Following TORS — Shortened Course Adjuvant Radiotherapy Following TORS

SUMMARY:
This is a single-arm, phase II study to establish the safety of reducing radiation dose in selected HPV-Associated OPSCC patients receiving adjuvant radiation after TORS and neck dissection. This protocol also allows for sparing of the primary resection bed, in appropriate patients, as previously published by our group and found to be safe and effective.

DETAILED DESCRIPTION:
This is a single-arm Phase II non-inferiority study of adjuvant radiation for locally-advanced HPV-Associated oropharyngeal squamous cell carcinoma. Patients with pT0-T3, N0-N1, M0 disease (per AJCC 8th Edition), detectable pre-operative and undetectable postoperative ctHPVDNA will be eligible. Patients will have undergone TORS primary site resection and neck dissection. Patients will undergo adjuvant RT +/- guideline-indicated chemotherapy. The neck and the primary site will be considered separately.

The primary objective of the study will be to determine the 2-year locoregional control (LRC) rate. Secondary objectives include measures of toxicity (as measured by CTCAE, version 5.0), patient-reported QOL (as measured by the MDASI and MDADI questionnaire), progression-free survival, metastasis-free survival, and overall survival. Differences between patients treated with IMRT and proton therapy in terms of toxicity and QOL will serve as another secondary objective.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Histologically confirmed diagnosis of squamous cell carcinoma of the oropharynx, p16-positive on immunohistochemistry or HPV-positive by In-Situ Hybridization
* Pathologic T0 (unknown primary), T1, T2, or T3 disease (per AJCC 8th Ed)
* Pathologic N0-N1 disease (per AJCC 8th Ed)
* Preoperative plasma ctHPVDNA of ≥ 50 copies/mL
* Undetectable postoperative plasma ctHPVDNA
* ECOG Performance Status 0-1

Exclusion Criteria:

* Prior external beam radiation therapy to the head and neck
* Presence of T4 disease
* ≥ 5 positive lymph nodes (which is pathologic N2 disease, per AJCC 8th edition)
* Presence of distant metastatic disease
* Uncontrolled inter-current illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, connective tissue disease or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Locoregional control | 2 years
  To determine whether disease recurs locally (at primary site) or in regionally in the nodes of the neck

SECONDARY OUTCOMES:
Progression-free survival | 2 Years
  To determine progression-free survival (any progression)
Metastasis-free survival | 2 years
  To determine metastasis-free survival (any distant metastasis)
Overall survival | 2 years
  To determine overall survival (alive or not)
Differences in toxicity between patients receiving IMRT and patients receiving PBT | 2 years
  To assess toxicity using the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Patient-Reported Quality of Life using MDASI-HN | 2 years
  The MD Anderson Symptom Inventory - Head & Neck (MDASI-HN)
  1. Minimum Value: 0
  2. Maximum Value: 280
  3. Higher scores mean worse outcome
Patient-Reported Quality of Life using MDADI | 2 years
  The MD Anderson Dysphagia Inventory (MDADI)
  1. Minimum Value: 20
  2. Maximum Value: 100
  3. Higher scores mean better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Lin, MD, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No